CLINICAL TRIAL: NCT07274618
Title: "Group Based Reverse OSCE" for Teaching Mechanical Ventilation to Nursing Students: A Randomized Controlled Trial
Brief Title: "Group Based Reverse OSCE" for Teaching Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Torbat Heydariyeh University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Alireza Sardashti, Director of program, Torbat Heydariyeh University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 402000038
Record Dates: First submitted 2025-11-26; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Medical Education; Nursing Students
Keywords: Simulation-based education; Mechanical ventilation training; Reverse OSCE; Competency-based medical education; Nursing students
MeSH Terms: interventions — Respiration, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- control group (Other): traditional method of education is being provided in this group
  Interventions: Other: mechanical ventilation (MV)

INTERVENTIONS:
Other: mechanical ventilation (MV) — in this educational intervention, nursing students are allocated to the reverse OSCE group in which the OSCE is being used for teaching mechanical ventilation education instead of acquiring test from student.

SUMMARY:
Introduction: Mechanical ventilation (MV) is a critical skill for healthcare professionals, yet traditional teaching methods often fail to adequately prepare students. This study evaluates the effectiveness of an innovative Group-Based Reverse OSCE.

Methods: A quasi-experimental study was conducted with 70 nursing students randomly assigned to either the Reverse OSCE group (n=35) or traditional lecture-based group (n=35). The intervention consisted of a 10-hour workshop featuring five interactive OSCE stations covering ventilator hardware, settings, modes, and alarm management. Knowledge and skills were assessed using validated pre- and post-tests, with statistical analysis performed via independent and paired t-tests (SPSS v25).

ELIGIBILITY:
Inclusion Criteria:

students from the nursing discipline who were in their clinical internship or clerkship students who completed relevant coursework in respiratory physiology, and had successfully passed the theoretical course in critical care.

no prior participation in similar ventilator training workshops within the past six months, demonstrating willingness for voluntary participation, and being able to attend the full 10-hour workshop (including both theoretical and practical components).

Exclusion Criteria:

partial attendance in the workshop, withdrawal at any stage of the study the occurrence of acute medical or emergency conditions interfering with participation or failure to complete the pre- and post-intervention assessment tools.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Mechanical ventilation knowledge | 1 day
  To assess students' knowledge and clinical reasoning in mechanical ventilation, a researcher-developed, mixed-format questionnaire was used. The tool included 20 items such as multiple-choice questions, clinical scenarios, calculation-based items (e.g., RSBI, ventilator settings), and graphic interpretation tasks. Content areas covered ventilator modes, complications, alarm settings, ABG analysis, and weaning criteria, designed in alignment with recent guidelines including the American Heart Association (2023).

CONTACTS AND LOCATIONS:
Locations (1):
- Torbat-e Heydariyeh University of Medical Sciences, Torbat-e Ḩeydarīyeh, Iran

IPD SHARING:
Plan to Share IPD: No
This study has been conducted on nursing student and confidentiality of data was promised to participants before this study began